CLINICAL TRIAL: NCT00326352
Title: Comparison of Sedation/Analgesia: Midazolam/Morphine Vs Propofol/Remifentanil
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003/1/13
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2006-05-16 (Estimated); Status verified 2006-05

CONDITIONS: Shoulder Dislocation
Keywords: Sedation; Propofol; Remifentanil; recovery
MeSH Terms: conditions — Shoulder Dislocation | interventions — Propofol; Remifentanil

INTERVENTIONS:
Drug: Sedation with propofol and remifentanil

SUMMARY:
For reduction of dislocated shoulder, sedation with propofol and remifentanil should give satisfactory operating conditions and pain relief, and significantly reduce the time to full recovery, compared with morphine and midazolam

DETAILED DESCRIPTION:
Propofol is a recognised agent for sedation and remifentanil is a short acting opioid analgesic. We intend to provide sedation with propofol, 0.5 mg/Kg, and analgesia with remifentanil 0.5 microgram/Kg for reduction of dislocated shoulders. This will be a randomised sex-stratified comparison with current therapy which is midazolam incrementally up to a maximum of 0.15 mg/Kg, and morphine incrementally up to 0.15 mg/Kg. The primary outcome measure is time to full recovery. Secondary aspects are pain or discomfort during the procedure and operating conditions.

ELIGIBILITY:
Inclusion Criteria:

- Anterior dislocation of the shoulder suitable for manual reduction

Exclusion Criteria:

* significant other illness
* body weight 25% greater than expected
* fear of oxygen masks
* alcohol intoxication

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-07; Study Completion 2005-06

PRIMARY OUTCOMES:
Time to full recovery

SECONDARY OUTCOMES:
Operating conditions
Pain or discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Gordon B Drummond, FRCA, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Background] Dunn MJ, Mitchell R, Souza CD, Drummond G. Evaluation of propofol and remifentanil for intravenous sedation for reducing shoulder dislocations in the emergency department. Emerg Med J. 2006 Jan;23(1):57-8. doi: 10.1136/emj.2004.021410. PMID 16373806